CLINICAL TRIAL: NCT02845739
Title: Study of the Distribution of Genotypes of HPV at the Ano-genital Area and Peripheral Humoral Immune Response Before and After Kidney Transplantation
Brief Title: PApillomavirus in REnal Transplant Patient
Acronym: PATRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: API/2009/09
Record Dates: First submitted 2016-07-12; First posted 2016-07-27 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Papillomavirus Infections
Keywords: kidney transplantation; human papillomavirus
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- kidney transplanted patient (Experimental)
  Interventions: Other: Kidney transplanted patients

INTERVENTIONS:
Other: Kidney transplanted patients

SUMMARY:
The main goal of project is to study the distribution of HPV genotypes in the anogenital area and peripheral humoral immune responses HPV (total and neutralizing Ab) before and after renal transplantation. Furthermore, the investigators wish (i) establish whether there is a correlation between HPV infection and HPV immune response before and after transplantation, and (ii) determine whether there is a link between HPV infection and immunosuppression.

DETAILED DESCRIPTION:
Kidney transplant patients, iatrogenic immunosuppression established, essential to limit the transplant. Kidney transplant patients, iatrogenic immunosuppression established, essential to limit the transplant rejection, exposes patients to an increased risk of infections, including human papillomavirus (HPV).

These patients thus constitute a population at risk of developing cancers associated with HPV. Indeed, a recent meta-analysis indicated that the standardized incidence ratio for cancers associated with HPV increases dramatically in kidney transplant: SIR of 2.13 (95% CI 1.37 to 3.30) for the cervical, RIS 22.76 (95% CI 15.8 to 32.7) for the vulva and vagina, RIS 15.8 (95% CI 5.79 to 34.40) for the penis, RIS 4.85 (95% CI 1.36 to 17.3) and RIS to the anus of 3.23 (95% CI 2.40 to 4.35) for the oral cavity and pharynx. In fact, transplant patients are subject to increased surveillance to detect the onset and / or progression of lesions (pre) cancerous, especially anogenital level. Data on HPV infection in the genital area of kidney transplant patients are few and concern cohorts with a modest number of subjects. Indeed, it is difficult to estimate the prevalence of infection and know precisely genotypes of HPV present in anogenital level. Similarly, some studies report the presence of anti-HPV antibodies in transplant patients.

The main goal of project is to study the distribution of HPV genotypes in the anogenital area and peripheral humoral immune responses HPV (total and neutralizing Ab) before and after renal transplantation. Furthermore, the investigators wish (i) establish whether there is a correlation between HPV infection and HPV immune response before and after transplantation, and (ii) determine whether there is a link between HPV infection and immunosuppression.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged over 18 years
* Patient waiting for first kidney transplant
* Patients receiving a social security scheme
* Postmenopausal women, surgically sterile or subjected to an effective method of contraception
* Patient who signed the written consent

Exclusion Criteria:

* Patients who have been transplanted
* Pregnant women
* Emergency situation Patients
* Patients unable to give consent personally
* Major protected Patients
* Patients under judicial supervision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2017-11-10 (Actual); Study Completion 2017-11-10 (Actual)

PRIMARY OUTCOMES:
Prevalence of genital HPV infection before and after kidney transplantation in man and women | 12 months
  For woman, gynecologist perform cervical and anal samples with DNA pap cervical sampler.
  For men, dermatologist perform penis and anal samples with same device. The sample with perform when the patient are registered to waiting list for transplant and 3 months and one year after transplantation.
  The samples are genotyped using the kit INNO-LiPA HPV Genotyping Extra test (Innogenetics) which allows the detection of 28 HPV types.

SECONDARY OUTCOMES:
Anti-HPV 16 Antibody titer in blood before and after kidney transplantation in man and women | 12 months
  Blood sample are taken in patient before, the day of transplantation and before. Titer (UI) of anti-HPV 16 antibody a serology is performed by ELISA.
Anti-HPV 18 Antibody titer in blood before and after kidney transplantation in man | 12 months
  Blood sample are taken in patient before, the day of transplantation and before. Titer (UI) of anti-HPV 18 antibody a serology is performed by ELISA.

IPD SHARING:
Plan to Share IPD: No